CLINICAL TRIAL: NCT03728517
Title: Comparison of Inpatient Narcotics Use to Outpatient Prescription Narcotics Post-operatively
Brief Title: Narcotics Inpatient / Outpatient
Status: Terminated | Type: Observational
Why Stopped: Low recruitment
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Insiyyah Patanwala, Principle Investigator, Indiana University
Other Study IDs: 1805708779
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Narcotic Use
Keywords: Narcotic; Inpatient; Outpatient; Comparison

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects who undergo gynecologic surgery: Subjects who will undergo gynecologic surgery via vaginally, laparoscopic , or robotic who require observation or inpatient stay overnight. This group will receive pain medication in the hospital and will also be discharged home with pain medication.

SUMMARY:
Managing pain in postoperative patients presents challenges in striking a balance between achieving adequate pain control and over-prescribing opioids that have the potential to contribute to the opioid epidemic. There are no clear guidelines informing postoperative opioid prescribing in obstetrics and gynecology.

The primary aim for this study are to better understand the factors that impact opioid use for pain management in gynecologic surgery patient after discharge. The second aim is to develop a model that incorporates individual patient baseline measures (e.g. anxiety, fibromyalgia score, inpatient narcotic consumption) to predict the amount of opioids needed following discharge.

DETAILED DESCRIPTION:
Managing pain in postoperative patients presents challenges in striking a balance between achieving adequate pain control and over-prescribing opioids that have the potential to contribute to the opioid epidemic. There are no clear guidelines informing postoperative opioid prescribing in obstetrics and gynecology. A recent study by As-Sanie et al. demonstrated that gynecologists at a large academic medical center prescribe twice the amount of opioids than the average patient uses after hysterectomy.1 Similarly, a study completed at Vanderbilt University Medical Center showed that obstetricians were overprescribing narcotics to patients after cesarean deliveries.2

In addition to rates of opioid prescribing, other factors affect postoperative opioid consumption, including individual patient measures of anxiety, depression, and self-reported pain scores prior to surgery. Preoperative Fibromyalgia symptom scores, STAIT state anxiety scores and NRS pain expectations are independent predictors for morphine consumption following hysterectomy.

There is a pressing need to better understand the factors that impact opioid use in women who undergo gynecologic surgery in order to mitigate the over-use of opioids for pain control upon discharge from the hospital.

Aims:

1. Understand the factors that impact opioid use for pain management in gynecologic surgery patients after discharge.

   1. Is opioid consumption during the immediate postoperative recovery phase associated with consumption after discharge?
   2. Are variables that are known to be associated with opioid consumption, also associated with opioid consumption after discharge?
   3. Are there factors which we can use to predict opioid consumption in postoperative patients?
2. Develop a model that incorporates individual patient baseline measures (e.g. anxiety, fibromyalgia score, inpatient narcotic consumption) to predict the amount of opioids needed following discharge.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Undergoing vaginal, laparoscopic or robotic gynecologic surgery requiring observation or inpatient stay overnight
* Agree to receiving contact from research staff for follow up
* Can provide two telephone numbers or a telephone number and email address

Exclusion Criteria:

* Unable to provide informed consent
* Age <18
* Intolerance/allergy to more than two narcotic medications
* Allergy/contraindication to non-steroidal anti-inflammatory drugs (NSAIDs)
* Has a diagnosed gynecologic malignancy other than Grade 1 endometrial cancer
* Pregnant
* Current opioid use on a regular basis (more than twice per week)
* Illicit drug-use within the past 30 days

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Subjects who are 18 years old or older who will have a vaginal , laparoscopic, or robotic surgery who require observation of an inpatient stay post-operatively.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Understand the factors that impact opioid use for pain management in gynecologic surgery patients after discharge. | 1 year
  1. Is opioid consumption during the immediate postoperative recovery phase associated with consumption after discharge?
  2. Are variables that are known to be associated with opioid consumption, also associated with opioid consumption after discharge?
  3. Are there factors which we can use to predict opioid consumption in postoperative patients?

SECONDARY OUTCOMES:
Develop a model | 1 year
  2. Develop a model that incorporates individual patient baseline measures (e.g. anxiety, fibromyalgia score, inpatient narcotic consumption) to predict the amount of opioids needed following discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Insiyyah Y Patanwala, Principal Investigator — Indiana School of Medicine
Locations (3):
- United States (3):
  - Eskenazi Health Hospital, Indianapolis, Indiana
  - Indiana University, Indianapolis, Indiana
  - Methodist Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Undecided